CLINICAL TRIAL: NCT05389748
Title: Phase IIb to Restore Oxygen in Large Vessel Occlusion Patients En Route for MT Using NanO2
Brief Title: NanO2 for Large Vessel Occlusion Stroke
Acronym: PROVEN
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NuvOx LLC (Industry)
Collaborators: University of Arkansas (Other); Stanford University (Other); Washington Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROVEN-P2
Record Dates: First submitted 2022-05-17; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Stroke
Keywords: perfusion; penumbra; mechanical thrombectomy; large vessel occlusion stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo which appears the same as the treatment to investigators, clinicians and subjects.
  Interventions: Other: Placebo
- NanO2 (Active Comparator): A milky white intravenous injectable emulsion
  Interventions: Biological: dodecafluoropentane emulsion (DDFPe)

INTERVENTIONS:
Other: Placebo — Subjects with large vessel occlusion stroke eligible for mechanical thrombectomy are randomized to placebo in association with standard of care
  Arms: Placebo
Biological: dodecafluoropentane emulsion (DDFPe) — Subjects with large vessel occlusion stroke eligible for mechanical thrombectomy are randomized to DDFPe in association with standard of care
  Arms: NanO2

SUMMARY:
A two stage phase 2 study with an interim analysis to provide evidence that subjects provided with early administration of NanO2 who are located at small rural spoke hospitals and identified with large vessel occlusion ischemic strokes as well as viable penumbra prior to transfer to larger hub hospitals and who continue dosing NanO2 until revascularization is achieved by intravenous alteplase and/or mechanical thrombectomy, will experience stroke recovery by shifting ischemic brain tissue to normal tissue pO2 environments.

DETAILED DESCRIPTION:
Recent stroke studies have shown that subjects with Large Vessel Occlusion (LVO) ischemic stroke have rapid infarct growth. The investigators hypothesize that early administration of NanO2 in subjects with LVO ischemic stroke will maintain the viability of tissue in the penumbra until revascularization is achieved with intravenous alteplase and/or mechanical thrombectomy (MT).

The rationale for administering the dose evaluated is:

1. The dose level is within the levels already tested in animals and humans.5-13 Volunteers received two IV bolus doses of 0.35 mL/kg of activated NanO2TM 24 hours apart and brain cancer subjects received daily doses of up to 0.17 mL/kg of inactivated NanO2TM.18
2. A completed trial of NanO2TM in acute ischemic stroke at the University of Arkansas had the high dose cohort receive three doses of NanO2 (0.17 mL/kg) 90 minutes apart and demonstrated safety at this dose.
3. Therapeutic reduction in stroke damage has been observed at dose levels of 0.1 mL/kg in rabbits.5-9,12 Since drug effects tend to correlate with body surface area/weight, one would predict that a dose of approximately 0.03 mL/kg should be effective in humans compared to rabbits.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 90 years old, male or female
* Diagnosis of LVO ischemic stroke
* Pre-stroke mRS ≤ 2
* NIHSS ≥ 6
* Eligible for mechanical thrombectomy per local criteria
* Subject or LAR must be willing and able to understand the study and provide written informed consent
* Women of childbearing potential or men with child-bearing potential partners (unless vasectomized) must agree to use a highly effective method of birth control from study entry until 4 months after completing study therapy. Should a study participant or their partner become pregnant or suspect a pregnancy they should inform the treating study physician immediately

Exclusion Criteria:

* > 12 hours since onset of stroke symptoms
* Currently pregnant or breastfeeding
* History of significantly impaired renal or hepatic function
* Severe hemorrhage or severe hemorrhagic stroke on CT scan. Mild or moderate changes of Fisher Grade 1 or 2 subarachnoid hemorrhage are allowed as are hemorrhagic transformation changes of Grade HI-1 and HI-224,25
* Unable to undergo a contrast brain perfusion scan with either MRI or CT
* Pre-stroke mRS > 2 (See Appendix 3)
* Unstable angina, NYHA Class II or greater congestive heart failure
* Uncontrolled hypertension (Systolic BP ≥ 200 and/or Diastolic BP ≤ 120 mmHg)
* Uncontrolled arrhythmia or history of clinically significant arrhythmia within the past six (6) months (except atrial fibrillation)
* Current acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy.
* History of allergic reaction attributed to compounds of similar chemical composition to NanO2TM (see Investigator's Brochure).
* Subject has received any investigational drug within thirty (30) days prior to enrollment into the study
* Inability to comply with the study procedures
* History or evidence of any other clinically significant condition that, in the opinion of the investigator, might pose a safety risk to subjects or interfere with study procedures, evaluation, or completion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale and Modified Rankin Scale | 2 years
  Both are established and accepted measures of stroke. NIHSS has a scale from 0 to 42 and mRS has a scale from 0 to 6. In both cases, a lower score represents less brain damage.